CLINICAL TRIAL: NCT05557019
Title: Semi Occlusion of the Coronary Sinus as an Adjunct to PCI in STEMI Patients, FIH Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intratech Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-002
Record Dates: First submitted 2022-09-18; First posted 2022-09-27 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Booster Balloon Therapy (Experimental): The Booster balloon therapy (i.e. partial occlusion of the CS lumen with a subsequent backward pressure elevation without obstructing the CS blood flow) will start immediately after a successful PCI of the culprit coronary lesion in the LAD, with TIMI-II flow restoration. The Booster balloon therapy will then be continued for up to 90 min, but not less than 60 min.
  Interventions: Device: Booster Balloon Catheter

INTERVENTIONS:
Device: Booster Balloon Catheter — The Booster balloon therapy (i.e. partial occlusion of the CS lumen with a subsequent backward pressure elevation without obstructing the CS blood flow) will start immediately after a successful PCI of the culprit coronary lesion in the LAD, with TIMI-II flow restoration. The Booster balloon therapy will then be continued for up to 90 min, but not less than 60 min.

SUMMARY:
The present study is planned to evaluate the safety and feasibility of the Booster Balloon catheter when applied to STEMI patients. The Booster Balloon is a spiral balloon intended to be positioned in the coronary sinus, enabling continuous venous draining while reducing flow and increasing the pressure inside the venous capillaries, and redistributing blood and oxygen to the border zone of the ischemic myocardium. This pilot, first-in-human study is designed to evaluate (in addition to safety and feasibility) the treatment modality in the setting of acute STEMI, as adjunctive therapy after restoring blood blow through the infract-related artery.

DETAILED DESCRIPTION:
The Booster Balloon Catheter, while inflated, causes partial occlusion of CS blood flow and thus increases the coronary sinus venous pressure. It is hypothesized that the utilization of a long pressure plateau, without a complete occlusion of the CS, will enable prolonged and improved redistribution of the venous flow and improve the oxygenation of the border zone (penumbra) of the infarcted myocardium at risk. The improved oxygenation of the ischemic peri-infarcted area is believed to reduce infarct size and may lead to improved short- and long-term outcomes.

This is a First-In-Human study aimed to evaluate the safety and feasibility of the Booster Balloon Catheter (BBC). The study will include up to 20 patients in up to 5 centers in Israel and Europe.

After the patients sign the informed consent, all the eligibility criteria will be evaluated. If a subject is found to be ineligible, the subject will be considered a "screen failure". Subjects who meet eligibility criteria will be treated with the BBC.

The total duration of subject participation will be 30±7 days.

ELIGIBILITY:
Inclusion Criteria:

Pre procedural:

1. Age above 18 years of age
2. Clinical presentation of anterior wall STEMI (ST-segment elevation > 1 mm in two or more contiguous leads between V1 and V4 or new left bundle branch block (LBBB)
3. STEMI culprit lesion in LAD
4. < 24-hour duration from time of symptom onset until admission to the emergency room
5. Patient providing informed consent compatible with the requirement of the institutional ethical committee.
6. Patient and physician agree to all required follow-up procedures and visits

   Angiographic inclusion criteria:
7. Coronary sinus diameter of 10 mm
8. PCI is indicated for culprit lesion in the LAD with planned use of a stent
9. Initial recanalization is successful, defined by stable culprit lesion and ≥ TIMI-2 flow and no major complications (detailed below).

Exclusion Criteria:

Pre-Procedure

1. Previous coronary artery bypass graft surgery
2. Previous anterior wall MI
3. Electrophysiology electrode in the coronary sinus (ICD, CRT)
4. History of stroke, transient ischemic attack, or any reversible ischemic neurological disease within the last 6 months
5. Pre-MI symptoms of CHF or known LVEF of <30%
6. Pre-MI-Known anemia (Hb <10).
7. Pre-MI Known severe renal failure (eGFR < 30 ml/min/1.73m2) or history of dialysis or renal transplant
8. Unconscious status
9. Contraindications to anticoagulant therapy, including hemorrhagic diathesis or thrombocytopenia
10. Pregnant women
11. Life expectancy < 1 year
12. Use of oral anticoagulant which is expected to be active at presentation.
13. Contraindications to adenosine
14. Hemodynamic instability, including pulmonary edema, cardiogenic shock
15. Current participation in other investigational device or drug trials that have not completed the primary efficacy endpoint follow-up parameters
16. Physician discretion that the patient should not be enrolled Intra-procedural
17. Coronary sinus anatomy which precludes patient from participation in the study
18. Hemodynamic instability, including cardiogenic shock or treatment with inotropes or vasopressors before, or during the PCI
19. Pulmonary edema
20. Acute complications of the MI
21. Complication of the PCI
22. Any medical condition that may be associated with a reduced prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events rate | 30 days
  Device or procedure related SAEs through hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Giora Weisz, MD, Study Director
Locations (2):
- Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi, Georgia
- Haemek Medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No